CLINICAL TRIAL: NCT06764108
Title: Multimodality Adaptive Intervention for Post-Inpatient Hospitalization Suicide Risk Reduction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rebecca G. Fortgang, Ph.D., Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R01MH139522 (NIH)
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Suicidal Ideation; Suicidal Behavior
Keywords: just-in-time adaptive intervention; JITAI; micro-randomized trial; MRT; Sequential Multiple Assignment Randomized Trial; SMART; single-session intervention; SSI; hybrid experimental design
MeSH Terms: conditions — Suicidal Ideation | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: This study uses a hybrid experimental design that embeds a Sequential Multiple Assignment Randomized Trial (SMART) and a Micro-Randomized Trial (MRT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Self-monitoring only (Experimental): Participants in the self-monitoring condition will complete smartphone-based self-monitoring of suicidal thoughts and related experiences during the four weeks after hospitalization. Those who exhibit a response to self-monitoring alone will not receive any add-on interventions.
  Interventions: Behavioral: Self-monitoring
- Self-monitoring plus JITAI (Experimental): Participants in the self-monitoring plus just-in-time adaptive intervention (JITAI) condition will complete smartphone-based self-monitoring of suicidal thoughts and related experiences during the four weeks after hospitalization. When they report experiencing suicidal thoughts on a self-monitoring survey, they may be randomly assigned to receive a JITAI comprising a brief series of automated smartphone-based messages recommending coping strategies for suicidal thoughts. Those who exhibit a response to self-monitoring plus JITAI will not receive any add-on interventions.
  Interventions: Behavioral: Self-monitoring; Behavioral: JITAI
- Self-monitoring only plus self-guided SSI (Experimental): Participants who are initially assigned to self-monitoring alone and do not sufficiently respond to this intervention (based on the previous week of self-monitoring data) may be randomly assigned to receive up to three brief online self-guided single-session interventions (SSIs) aimed to identify and address barriers to coping strategy use during the four weeks after hospitalization.
  Interventions: Behavioral: Self-monitoring; Behavioral: Self-guided SSI
- Self-monitoring only plus clinician-delivered SSI (Experimental): Participants who are initially assigned to self-monitoring alone and do not sufficiently respond to this intervention (based on the previous week of self-monitoring data) may be randomly assigned to receive up to three single-session interventions (SSIs) with a study clinician aimed to identify and address barriers to coping strategy use during the four weeks after hospitalization.
  Interventions: Behavioral: Self-monitoring; Behavioral: Clinician-delivered SSI
- Self-monitoring plus JITAI plus self-guided SSI (Experimental): Participants who are initially assigned to self-monitoring plus JITAI and do not sufficiently respond to this intervention (based on the previous week of self-monitoring data) may be randomly assigned to receive up to three brief online self-guided SSIs aimed to identify and address barriers to coping strategy use during the four weeks after hospitalization.
  Interventions: Behavioral: Self-monitoring; Behavioral: JITAI; Behavioral: Self-guided SSI
- Self-monitoring plus JITAI plus clinician-delivered SSI (Experimental): Participants who are initially assigned to self-monitoring plus JITAI and do not sufficiently respond to this intervention (based on the previous week of self-monitoring data) may be randomly assigned to receive up to three sessions with a study clinician aimed to identify and address barriers to coping strategy use during the four weeks after hospitalization.
  Interventions: Behavioral: Self-monitoring; Behavioral: JITAI; Behavioral: Clinician-delivered SSI

INTERVENTIONS:
Behavioral: Self-monitoring — Self-monitoring will involve completing one brief smartphone-based survey (at a fixed time) per day on suicidal thoughts and related affect states and experiences over the past day during the four weeks after psychiatric hospitalization.
Behavioral: JITAI — The JITAI will involve prompts to complete additional randomly timed self-monitoring surveys throughout the day. When suicidal thoughts are reported on any self-monitoring survey, random assignment to receive or not receive a series of automated smartphone-based messages that recommend using specific coping strategies from either a personalized safety plan or general evidence-based coping strategies that others tend to find helpful.
  Arms: Self-monitoring plus JITAI; Self-monitoring plus JITAI plus clinician-delivered SSI; Self-monitoring plus JITAI plus self-guided SSI
Behavioral: Self-guided SSI — The brief (10-12 minute) online self-guided SSI will help individuals identify and address barriers to using coping strategies for suicidal thoughts. It may be delivered up to three times during the four weeks after hospitalization for those who do not sufficiently respond to the initial (self-monitoring only or self-monitoring plus JITAI) interventions.
  Arms: Self-monitoring only plus self-guided SSI; Self-monitoring plus JITAI plus self-guided SSI
Behavioral: Clinician-delivered SSI — The clinician-delivered SSI will consist of a brief (30-minute) Zoom or phone meeting in which a study clinician will help individuals identify and address barriers to using coping strategies for suicidal thoughts. Those who do not sufficiently respond to the initial (self-monitoring only or self-monitoring plus JITAI) interventions may receive up to three clinician-delivered SSIs during the four weeks after hospitalization.
  Arms: Self-monitoring only plus clinician-delivered SSI; Self-monitoring plus JITAI plus clinician-delivered SSI

SUMMARY:
The goal of this clinical trial is to learn whether a combination of brief digital and clinician-delivered interventions can help adults leaving a psychiatric hospitalization cope with suicidal thoughts and prevent suicide-related events.

The main questions it aims to answer are:

* Are people who receive automated smartphone messages when they report suicidal thoughts after leaving the hospital less likely to have a suicide-related event than those who do smartphone self-monitoring alone?
* Are people who have additional session(s) with a clinician in the four weeks after leaving the hospital less likely to have a suicide-related event than those who receive additional brief self-guided intervention(s)?

Participants will be asked to:

* Make a personalized safety plan (of coping strategies to use when feeling suicidal) before leaving the hospital
* Do self-monitoring of suicidal thoughts and related experiences on their smartphone for four weeks after leaving the hospital
* Complete a longer set of research questionnaires at the start of the study and five more times during the 12 weeks after leaving the hospital

Depending on which study group they are in and whether they benefit from initial smartphone interventions, participants may or may not:

* Receive automated smartphone messages reminding them of coping strategies to use for suicidal thoughts
* Receive up to three additional sessions with a study clinician
* Receive up to three brief online self-guided interventions

The study interventions last for the four weeks after leaving the hospital. Participants will also be asked permission to share information from their health records about care received for 12 weeks after leaving the hospital.

DETAILED DESCRIPTION:
Over 49,000 Americans die by suicide each year, making suicide the 11th leading cause of death across all ages. The highest-risk time for suicidal behavior is the three months after inpatient psychiatric hospitalization, during which engagement with traditional outpatient care is low. Recent real-time monitoring research has revealed that suicidal thoughts fluctuate rapidly, over hours or even minutes, highlighting the need for dynamic interventions that adapt to time-varying changes in risk. Just-in-time adaptive interventions (JITAIs) can help promote timely coping strategy use during periods of elevated suicidal thinking. Some people, however, will require additional interventions that explicitly target common barriers to coping effectively with suicidal thoughts. Evidence-based single-session interventions (SSIs) that address coping with suicidal thoughts exist and can be delivered in either clinician-delivered or self-guided formats. This study will use a hybrid experimental design that leverages both Sequential Multiple Assignment Randomized Trial and Micro-Randomized Trial (MRT) methods to build and evaluate a multimodality adaptive intervention comprising stepped evidence-based intervention components sequenced and adapted at multiple timescales following inpatient hospitalization.

Aim 1 will compare two first-stage interventions: JITAI vs. self-monitoring alone for four weeks after inpatient discharge. The investigators will determine the effectiveness of the JITAI for reducing the risk of suicide-related events (SREs) over three months and whether the JITAI engages target mechanisms related to coping.

Aim 2 will compare two second-stage interventions for those who do not sufficiently respond to the first-stage interventions: clinician-delivered or self-guided SSIs targeting individualized barriers to coping strategy use. Response status will be assessed weekly for four weeks post-hospitalization. The investigators will determine the effectiveness of clinician-delivered vs. self-guided SSIs for reducing the risk of SREs among insufficient responders, as well as effect differences between embedded adaptive interventions among all participants.

Aim 3 will determine the within-person effects of just-in-time messages on proximal outcomes (next-hour coping strategy use and momentary suicidal thoughts) for participants in the JITAI condition. Just-in-time message effects will be evaluated when averaging across second-stage conditions and contrasting message and SSI types.

This study will result in a scalable and optimized stepped approach to reducing suicide risk during a key care transition period.

ELIGIBILITY:
Inclusion Criteria:

* Adult status (18+ years-old)
* Ownership of a smartphone (iOS or Android)
* Inpatient admission due to suicidal thoughts or suicide attempt

Exclusion Criteria:

- Presence of any factor that impairs an individual's ability to comprehend and effectively participate in the study, including an inability to speak or write English fluently, the presence of gross cognitive impairment due to florid psychosis, intellectual disability, dementia, acute intoxication, or the presence of extremely agitated or violent behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-09 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Suicide-related event (SRE) | From inpatient discharge to the end of the study intervention period at 4 weeks
  SRE defined as suicide attempt or emergency visit/re-hospitalization for suicide risk

SECONDARY OUTCOMES:
Suicide-related event (SRE) | From inpatient discharge to the end of the study at 12 weeks
  SRE defined as suicide attempt or emergency visit/re-hospitalization for suicide risk
Coping strategy use | From inpatient discharge to the end of the study intervention period at 4 weeks
  Past-day coping strategy use will be operationalized with a variable indicating the proportion of days with suicidal thoughts when coping strategies for suicidal thoughts were used
Coping self-efficacy | From inpatient discharge to the end of the study intervention period at 4 weeks
  Past-week coping self-efficacy will be operationalized with Suicide-Related Coping Scale total scores, which range from 0 to 68, with higher scores indicating better coping.
Coping strategy use | From inpatient discharge to the end of the study intervention period at 4 weeks
  Coping strategy use since the last self-monitoring survey will be operationalized with a binary variable indicating whether evidence-based coping strategies were used to manage suicidal thoughts since the last survey.
Suicide urge intensity | MomentFrom inpatient discharge to the end of the study intervention period at 4 weeksary
  Momentary (current) suicide urge intensity will be rated on a 0 (not at all) - 10 (very strong) scale.
Suicide intent intensity | From inpatient discharge to the end of the study intervention period at 4 weeks
  Momentary (current) suicide intent intensity will be rated on a 0 - 10 scale.

IPD SHARING:
Plan to Share IPD: Yes
In accordance with NIH guidelines, individual participant data collected in this study (including self-report and demographic data), as well as a corresponding data dictionary, will be shared via the National Institute of Mental Health National Data Archive (NDA).